CLINICAL TRIAL: NCT06466720
Title: Measuring and Mapping Cognitive Decline After Brain Radiosurgery: a Pilot Study
Brief Title: Measuring and Mapping Cognitive Decline After Brain Radiosurgery
Acronym: CoDeB-Rad
Status: Recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 24016
Record Dates: First submitted 2024-06-04; First posted 2024-06-20 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-05

CONDITIONS: Brain Metastases; Meningiomas; Stereotactic Radiosurgery; Cognitive Decline; Quality of Life; SRS
Keywords: Brain metastases; Meningiomas; Stereotactic Radiosurgery; SRS; Cognitive Decline; Quality of Life
MeSH Terms: conditions — Brain Neoplasms; Meningioma; Cognitive Dysfunction | interventions — Mental Status and Dementia Tests; Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prospective: Patients with brain metastases and meningiomas that are eligible for SRS treatment will be included in the prospective arm of the trial. The patients will have neurocognitive testing in the form of the Montreal Cognitive Assessment (MoCA) and will answer two Quality of Life questionnaires (QLQs) by EORTC QLQ-C30 and BN20). The baseline visit will happen before they start their SRS treatment.
  The patients will be seen an additional 4 times, at 3, 6, 9 and 12 months after radiotherapy treatment. During each visit they will complete the MoCA and the QLQs.
  During the first follow up appointment they will also be asked to think back to before they had the treatment and answer the QLQs based on that.
  Interventions: Behavioral: Neurocognitive testing; Behavioral: Quality of Life questionnaire; Radiation: Stereotactic radiosurgery
- Retrospective: Patients with meningiomas that have received SRS treatment more than a year ago will be included in the retrospective arm of the trial. The patients will have neurocognitive testing in the form of the Montreal Cognitive Assessment (MoCA) and will answer two Quality of Life questionnaires (QLQs) by EORTC QLQ-C30 and BN20) once. They will also be asked to think back to before they had the treatment and answer the QLQs based on that.
  Interventions: Behavioral: Neurocognitive testing; Behavioral: Quality of Life questionnaire; Radiation: Stereotactic radiosurgery

INTERVENTIONS:
Behavioral: Neurocognitive testing — The MoCA is a brief tool developed to screen mild cognitive impairment and has been validated in patients aged 55-85 years old. It has been tested and validated in patients with brain metastases, and its acceptability has been tested in the general brain tumour population. The paper version of the MoCA is available in nearly 100 languages. The online version is available currently in 5 languages.
  Other Names: Montreal Cognitive Assessment
Behavioral: Quality of Life questionnaire — The EORTC-QLQ-C30 is a quality-of-life questionnaire that was developed by the European Organisation for Research and Treatment of Cancer (EORTC) for use in clinical trials. It is a 30-item questionnaire that incorporates the following five scales: physical, role, cognitive, emotional and social. It has also been validated and is available in more than 100 languages. The EORTC-QLQ-BN20 is a questionnaire that was developed for use specifically with patients that have brain cancer. The BN20 is a 20-item questionnaire and addresses four different scales (multi-item): future uncertainty, visual disorder, motor dysfunction and communication deficit. There are seven items that assess physical symptoms: headaches, seizures, drowsiness, hair loss, itchy skin, weakness of legs and bladder control. The questionnaire has been validated in over 15 languages. The two questionnaires are meant to complement each other when used in patients with brain cancer.
  Other Names: QLQ-C30; QLQ-BN20
Radiation: Stereotactic radiosurgery — This is a Standard of Care treatment for all the patients that will be recruited in both cohorts. Stereotactic radiosurgery will be delivered to one or more sites and in the prospective cohort can be delivered more than once.
  Other Names: SRS

SUMMARY:
Background Stereotactic Radiosurgery (SRS) is a localised radiotherapy treatment for patients with brain metastases or other benign tumours in the brain, like meningiomas. The Investigators do not currently know if, or how much, SRS affects brain function. Patients with brain tumours do not get tested routinely for their brain function.

Understanding short- and long-term side-effects is important for SRS. Brain metastases patients have short life expectancies (6-months to 1-year). However, meningioma patients can live 10 years or more. SRS is used to treat both.

The Montreal Cognitive Assessment will be used to test the participants' brain function. Quality-of-life questionnaires QLQ-C30 and BN20 will also be used to assess the participants' physical and mental wellbeing . These are specific for patients with brain cancer.

Why is it important This study aims to identify areas in the brain that relate to changes in brain function after SRS. These areas can then have the radiation dose reduced to them in future patients, hoping to minimise side-effects.

Research Question Which regions of the brain contribute to a decline in brain function following SRS.

Study Design This is a single centre observational study with prospective and retrospective collection of data.

This study will look at two groups of patients:

Group1: Patients will complete the MoCA and two quality-of-life questionnaires before the treatment and every 3 months for a year.

Group2: Patients will complete the MoCA and two quality-of-life questionnaires once.

The investigators will use these tests, MRI scans and the SRS treatment plan to identify areas of the brain that are responsible for any problems with the participants' brain function.

The participants for Group 1 will be recruited from the SRS Clinics, at City Campus, Nottingham University Hospitals NHS Trust.

The participants for Group 2 will be identified through the Mosaiq Oncology Information System.

This pilot study is funded by the Midlands Mental Health and Neurosciences Network.

DETAILED DESCRIPTION:
Brain metastases affect roughly 20-40% of all cancer patients with a primary extracranial disease. Lamba et at estimated that patients' median survival without treatment is approximately one month. This number increases from one month to between three and 12 months if whole brain radiotherapy (WBRT) is used. WBRT is a radiotherapy treatment that is delivered in five to ten sessions and where the whole brain is irradiated. With the advent of new systemic treatments, prognosis for patients is constantly improving . The widespread use of MRI imaging has also increased the number of patients being diagnosed by improving the detection of very small tumours (one or two millimetres in diameter). Consequently, more people are referred for treatment with a curative intent for their brain metastases.

Patients with brain metastases can be treated with surgery, WBRT, Stereotactic Radiosurgery (SRS) or a combination of the above. SRS is the treatment of choice for single or multiple metastases, unless there is a large mass (more than 3 cm in diameter) when surgery would be the preferred option. This is due to the invasiveness of the surgery, SRS is non or minimally invasive, and the associated risks of having a surgical resection. SRS is a highly focused treatment that makes use of stereotactic localisation techniques to deliver a high radiation dose to an outlined area of the brain. The treatment is usually delivered in a single radiotherapy treatment. In prospective randomised controlled trials, it was shown that Stereotactic Radiosurgery is as effective as whole brain radiotherapy, in terms of local tumour control, but the burden of cognitive decline for the patients is less. The primary tumours can vary, but the majority of the patients have a lung, breast, melanoma, kidney or colon primary.

Radiation damages the brain, with different areas being more or less susceptible to radiation. The main organs used to optimise radiotherapy treatment plans by reducing the dose delivered to these, include the eyes, optic nerves, chiasma, brainstem, cochleas, lenses and lacrimal glands. These are organs that affect physical functions. Currently, during radiotherapy treatment planning, no consideration is given to areas of the brain that affect cognitive function, such as the hippocampus, basal ganglia, insula and corpus callosum to name a few.

The effects of radiotherapy in the brain are well documented but this is mostly for WBRT. The effects of focal radiotherapy, such as SRS, on cognition have not been studied in detail. This pilot study will be using voxel-based lesion symptom mapping (VLSM) to correlate the treatment planning dose maps with clinical outcomes on neurocognitive function.

Voxel-based lesion symptom mapping is a technique where the relationship between damage to certain locations of the brain can be corelated with symptoms that affect cognitive function. This is done on a voxel-by-voxel basis. A voxel is a volume in a three-dimensional structure. VLSM has been used extensively in the past in stroke patients, but the literature is scarce for patients with brain metastases. Individual MR images of the brain will be used along with the dose maps from each patient's SRS treatment plan. The dose maps will be overlayed and correlated with results from neurocognitive testing. The identified areas of the brain will then be outlined and the dose level of significance (the level of dose at which cognitive change becomes quantifiable) will be assessed.

Benefits

The identification of areas in the brain and associated doses with cognitive changes will help advise future guidelines on volumetric dose constraints for those areas in the brain. As lesion location will be correlated with clinical outcomes from neurocognitive testing, a better understanding of the side-effects of the radiotherapy treatment may be gained. This will allow the optimisation of future radiotherapy treatments, to spare these areas thereby minimising the side-effects of the radiotherapy treatment.

Finally, with the acquired knowledge, consultants will be better placed to inform patients about the effects that their treatment will have. Patients will therefore be able to make informed decisions about their treatment. This is especially important in this population, as the majority of patients treated with SRS do not have a very long life-expectancy.

Methods Magnetic Resonance Imaging or MRI is a medical imaging technique that uses magnetic fields and radio waves to generate detailed images of the inside of the body. MRI is the preferred imaging method used to diagnose tumours in the brain, both benign and malignant, due to its ability to provide high contrast for these tissues. Tumours as small as 2 mm can be easily visualised with the aid of an MRI scanner.

The methodology that will be used to analyse the data, VLSM, is well established and has been used extensively in patients with stroke lesions. It uses a regression model that is univariate and can associate the cognitive performance of patients to whether or not a lesion is present in each voxel. In this pilot study instead of using lesions the investigators will be using the dose maps of the radiotherapy treatment plans.

The structural MRI scans of the patients will be spatially normalised to a common coordinate system, the Montreal Neurological Institute (MNI) space. The transformations will then be used to fit the dose maps to the same coordinate system. The data will then be smoothed. The voxel-based lesion symptom mapping analysis will involve the use of a Matlab statistical parametric mapping toolbox. For each voxel a group comparison between patients will be undertaken with the use of the dose maps from the radiotherapy treatment plans. The t statistic will be computed based on the results from the neurocognitive testing. A corresponding t-map of the brain will be created showing all the voxels related to the relevant cognitive deficits. A correction for multiple comparisons needs to be carried out to ensure that the rate of false positives will be minimised.

ELIGIBILITY:
Inclusion criteria Prospective Cohort

Patients will be eligible for inclusion only if ALL of the following criteria apply:

* Age: above 18 years, no upper limit
* Diagnosis of brain metastases or meningioma, where the treatment is going to be stereotactic radiosurgery
* Karnofsky Performance Status (KPS) ≥70
* Established diagnosis of cancer with absent or controllable primary disease
* Tumour volume of less than 20cc
* Life expectancy of more than 6 months
* Able to give informed consent

Exclusion criteria Prospective Cohort

* Previous RT to the brain, including SRS
* Previous surgery to the brain
* Not willing or not able to give informed consent

Inclusion criteria Retrospective Cohort

Patients will be eligible for inclusion only if ALL of the following criteria apply:

* Age: above 18 years, no upper limit
* Diagnosis of meningioma
* Previous SRS treatment at least 1 year prior to inclusion in the study
* Most recent MRI scan (within 1 year) shows stable appearances
* Able to give informed consent

Exclusion criteria Retrospective Cohort

* Previous RT to the brain, excluding SRS
* Previous surgery to the brain
* Not willing or not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is based within the East Midlands, United Kingdom. The East Midlands Stereotactic Radiosurgery (SRS) service covers Nottinghamshire, Derbyshire, Lincolnshire and Leicestershire. Any patients that are eligible for SRS (prospective cohort) or has already been treated with SRS (retrospective cohort) and also fulfil the eligibility criteria of the study will be invited to take part in the study.
  Patients will be recruited through the SRS clinics taking place at City Campus, Nottingham University Hospitals NHS Trust.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to neurocognitive function and Quality of Life at 6 months | 6 months
  Significant changes in neurocognitive function and Quality of Life at 6 months compared to baseline.The scale ranges from 0-100 with 0 signifying a worse quality of life and 100 signifying excellent quality of life for the participants. The cognitive function scale ranges from 0-30 with 30 signifying non-impaired cognitive function.
Doses related to neurocognitive symptoms | 6 months
  • Doses above which the lesion symptom mapping identifies areas of the brain relevant to neurocognitive symptoms at 6 months.

SECONDARY OUTCOMES:
Recruitment feasibility | 1.5 years
  The number of patients screened versus the number of patients recruited will be recorded along with any reasons for non-participation
Patient reported symptoms vs symptoms identified by neurocognitive testing | At baseline and every 3 months
  • Do patient reported symptoms relate to those identified from neurocognitive testing.

OTHER OUTCOMES:
Areas of the brain related to neurocognitive function | 6 months
  • Geographical correlation of areas in the brain with change in neurocognitive function as identified by Voxel based lesion symptom mapping
Identification of radiosensitive structures in the brain | 6 months
  • Identification of brain structures most affected by radiation via differences in the cognitive testing.

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Morgan, Professor of Medical Physics, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lamba N, Muskens IS, DiRisio AC, Meijer L, Briceno V, Edrees H, Aslam B, Minhas S, Verhoeff JJC, Kleynen CE, Smith TR, Mekary RA, Broekman ML. Stereotactic radiosurgery versus whole-brain radiotherapy after intracranial metastasis resection: a systematic review and meta-analysis. Radiat Oncol. 2017 Jun 24;12(1):106. doi: 10.1186/s13014-017-0840-x. PMID 28646895
- [Background] Lippitz B, Lindquist C, Paddick I, Peterson D, O'Neill K, Beaney R. Stereotactic radiosurgery in the treatment of brain metastases: the current evidence. Cancer Treat Rev. 2014 Feb;40(1):48-59. doi: 10.1016/j.ctrv.2013.05.002. Epub 2013 Jun 27. PMID 23810288
- [Background] Bates E, Wilson SM, Saygin AP, Dick F, Sereno MI, Knight RT, Dronkers NF. Voxel-based lesion-symptom mapping. Nat Neurosci. 2003 May;6(5):448-50. doi: 10.1038/nn1050. No abstract available. PMID 12704393
- [Background] Glascher J, Tranel D, Paul LK, Rudrauf D, Rorden C, Hornaday A, Grabowski T, Damasio H, Adolphs R. Lesion mapping of cognitive abilities linked to intelligence. Neuron. 2009 Mar 12;61(5):681-91. doi: 10.1016/j.neuron.2009.01.026. PMID 19285465
- [Background] Geva S, Baron JC, Jones PS, Price CJ, Warburton EA. A comparison of VLSM and VBM in a cohort of patients with post-stroke aphasia. Neuroimage Clin. 2012 Aug 30;1(1):37-47. doi: 10.1016/j.nicl.2012.08.003. eCollection 2012. PMID 24179735
- [Background] Taphoorn MJ, Claassens L, Aaronson NK, Coens C, Mauer M, Osoba D, Stupp R, Mirimanoff RO, van den Bent MJ, Bottomley A; EORTC Quality of Life Group, and Brain Cancer, NCIC and Radiotherapy Groups. An international validation study of the EORTC brain cancer module (EORTC QLQ-BN20) for assessing health-related quality of life and symptoms in brain cancer patients. Eur J Cancer. 2010 Apr;46(6):1033-40. doi: 10.1016/j.ejca.2010.01.012. Epub 2010 Feb 22. PMID 20181476
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Meyer S, Kessner SS, Cheng B, Bonstrup M, Schulz R, Hummel FC, De Bruyn N, Peeters A, Van Pesch V, Duprez T, Sunaert S, Schrooten M, Feys H, Gerloff C, Thomalla G, Thijs V, Verheyden G. Voxel-based lesion-symptom mapping of stroke lesions underlying somatosensory deficits. Neuroimage Clin. 2015 Dec 11;10:257-66. doi: 10.1016/j.nicl.2015.12.005. eCollection 2016. PMID 26900565
- [Background] Renovanz M, Reitzug L, Messing L, Scheurich A, Gruninger S, Ringel F, Coburger J. Patient reported feasibility and acceptance of Montreal Cognitive Assessment (MoCA) screening pre- and postoperatively in brain tumour patients. J Clin Neurosci. 2018 Jul;53:79-84. doi: 10.1016/j.jocn.2018.04.034. Epub 2018 Apr 20. PMID 29685411
- [Background] Olson RA, Iverson GL, Carolan H, Parkinson M, Brooks BL, McKenzie M. Prospective comparison of two cognitive screening tests: diagnostic accuracy and correlation with community integration and quality of life. J Neurooncol. 2011 Nov;105(2):337-44. doi: 10.1007/s11060-011-0595-4. Epub 2011 Apr 26. PMID 21520004
- [Background] Olson RA, Chhanabhai T, McKenzie M. Feasibility study of the Montreal Cognitive Assessment (MoCA) in patients with brain metastases. Support Care Cancer. 2008 Nov;16(11):1273-8. doi: 10.1007/s00520-008-0431-3. Epub 2008 Mar 12. PMID 18335256
- [Background] Yang Y, Tompkins CA, Meigh KM, Prat CS. Voxel-Based Lesion Symptom Mapping of Coarse Coding and Suppression Deficits in Patients With Right Hemisphere Damage. Am J Speech Lang Pathol. 2015 Nov;24(4):S939-52. doi: 10.1044/2015_AJSLP-14-0149. PMID 26425785
- [Background] Baldo JV, Schwartz S, Wilkins D, Dronkers NF. Role of frontal versus temporal cortex in verbal fluency as revealed by voxel-based lesion symptom mapping. J Int Neuropsychol Soc. 2006 Nov;12(6):896-900. doi: 10.1017/S1355617706061078. PMID 17064451
- [Background] DeMarco AT, Turkeltaub PE. A multivariate lesion symptom mapping toolbox and examination of lesion-volume biases and correction methods in lesion-symptom mapping. Hum Brain Mapp. 2018 Nov;39(11):4169-4182. doi: 10.1002/hbm.24289. Epub 2018 Jul 4. PMID 29972618
- [Background] Chang EL, Wefel JS, Hess KR, Allen PK, Lang FF, Kornguth DG, Arbuckle RB, Swint JM, Shiu AS, Maor MH, Meyers CA. Neurocognition in patients with brain metastases treated with radiosurgery or radiosurgery plus whole-brain irradiation: a randomised controlled trial. Lancet Oncol. 2009 Nov;10(11):1037-44. doi: 10.1016/S1470-2045(09)70263-3. Epub 2009 Oct 2. PMID 19801201
- [Background] Welzel G, Fleckenstein K, Mai SK, Hermann B, Kraus-Tiefenbacher U, Wenz F. Acute neurocognitive impairment during cranial radiation therapy in patients with intracranial tumors. Strahlenther Onkol. 2008 Dec;184(12):647-54. doi: 10.1007/s00066-008-1830-6. Epub 2008 Dec 24. PMID 19107345
- [Background] Lin X, DeAngelis LM. Treatment of Brain Metastases. J Clin Oncol. 2015 Oct 20;33(30):3475-84. doi: 10.1200/JCO.2015.60.9503. Epub 2015 Aug 17. PMID 26282648
- [Background] Tsao MN, Rades D, Wirth A, Lo SS, Danielson BL, Vichare A, Hahn C, Chang EL. International practice survey on the management of brain metastases: Third International Consensus Workshop on Palliative Radiotherapy and Symptom Control. Clin Oncol (R Coll Radiol). 2012 Aug;24(6):e81-92. doi: 10.1016/j.clon.2012.03.008. PMID 22794327
- [Background] Tsao MN, Xu W, Wong RK, Lloyd N, Laperriere N, Sahgal A, Rakovitch E, Chow E. Whole brain radiotherapy for the treatment of newly diagnosed multiple brain metastases. Cochrane Database Syst Rev. 2018 Jan 25;1(1):CD003869. doi: 10.1002/14651858.CD003869.pub4. PMID 29365347
- [Background] Brown PD, Jaeckle K, Ballman KV, Farace E, Cerhan JH, Anderson SK, Carrero XW, Barker FG 2nd, Deming R, Burri SH, Menard C, Chung C, Stieber VW, Pollock BE, Galanis E, Buckner JC, Asher AL. Effect of Radiosurgery Alone vs Radiosurgery With Whole Brain Radiation Therapy on Cognitive Function in Patients With 1 to 3 Brain Metastases: A Randomized Clinical Trial. JAMA. 2016 Jul 26;316(4):401-409. doi: 10.1001/jama.2016.9839. PMID 27458945
- [Derived] Bangiri A, Horobin A, Baker J, Pszczolkowski S, Thust S, Morgan PS. Outcomes of patient and public involvement in the development of the Cognitive Decline after Brain Radiosurgery (CoDe B-Rad) study: refining the research question and methodology. BMJ Open. 2025 Jun 26;15(6):e094788. doi: 10.1136/bmjopen-2024-094788. PMID 40578862
- See also: NHS Website, MRI Scan MRI scan - NHS (www.nhs.uk) , page last visited on 12/02/2024 — https://www.nhs.uk/conditions/mri-scan/